CLINICAL TRIAL: NCT02440399
Title: To Compare the Efficacy and Patients' Satisfaction for the Treatment of Post Cesarean Pain of Two Protocols: Oral Medications in Fixed Time Interval Administration Versus Spinal Morphine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, enav yefet, MD/PhD, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0028-15
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Post Cesarean Pain Management
MeSH Terms: interventions — Tramadol; Morphine; Acetaminophen; Diclofenac; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fix protocol - Oral treatment (Experimental): During 48 hours following surgery pain medications will be given as followed (listed in brackets are the generic names of each medication):
  At patient arrival to the department: Intravenous Tramadol hydrochloride 100 milligrams + TAB. Paracetamol 500 milligrams + TAB. Diclofenac 100 milligrams
  After 6 hours from patient arrival and every 6 hours: TAB. Zaldiar (Paracetamol 650 milligrams + Tramadol 75 milligrams).
  After 12, 24 and 48 hours from patient arrival: TAB. Diclofenac 100 milligrams.
  Rescue medication: TAB. Percocet (Oxycodone 5MG/Paracetamol 325 MG)as necessary up to 4 times per day.
  The total amount of paracetamol is limited to 4 gr per day.
  Interventions: Drug: Tramadol hydrochloride; Drug: Paracetamol; Drug: Diclofenac; Drug: TAB. Percocet (Oxycodone 5MG/Paracetamol 325 MG)
- Spinal morphine (Experimental): The women will receive 150 mcg morphine with the spinal anesthesia given in the cesarean section
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Tramadol hydrochloride — Please see arm description
  Arms: Fix protocol - Oral treatment
Drug: Morphine — Please see arm description
  Arms: Spinal morphine
Drug: Paracetamol
  Arms: Fix protocol - Oral treatment
Drug: Diclofenac
  Arms: Fix protocol - Oral treatment
Drug: TAB. Percocet (Oxycodone 5MG/Paracetamol 325 MG)
  Arms: Fix protocol - Oral treatment

SUMMARY:
Cesarean deliveries are prevalent. Unlike other operations, quick recovery is required for the mother to nurture the newborn child and establishing an appropriate mother-child bonding.

DETAILED DESCRIPTION:
Cesarean deliveries are prevalent. Unlike other operations, quick recovery is required for the mother to nurture the newborn child and establishing an appropriate mother-child bonding. Therefore, effective pain management is crucial. In this study we would like to compare between two pain relievers' administration protocols:

1. Oral pain relievers' administration in fix protocol without need for patient demand
2. Spinal morphine given during the spinal anesthesia in the cesarean section

ELIGIBILITY:
Inclusion Criteria:

* women that underwent cesarean section with sinal anesthesia

Exclusion Criteria:

* Women who suffer from chronic pain
* Women using chronic pain medications
* Women with allergy to any drug used in the study
* Women underwent general anesthesia during the surgery
* Women who suffer from sleep apnea
* Women who suffer from obesity (BMI>40)
* Women who suffer from severe nausea and vomiting after previous surgery
* Women who received perioperative magnesium
* Women who suffer from hypertension
* Women who suffer from renal failure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The efficacy of pain management | during 48 hours from surgery
  Pain sensation will be assessed using the NRS scale (numeric rating scale) for measurement of acute pain

SECONDARY OUTCOMES:
Patient satisfaction | 48 hours after surgery
  Each patient will fill in a satisfaction questioner which is given 48 hours after surgery
The necessity of additional medications (rescue doses) | During 48 hours after surgery
Adverse effect of the medications given in each protocol on the mother and neonates | during 48 hours following surgery
To compare the amount of breastfeeding between 2 groups | Following the week after surgery
Total amount of pain medications required in each study group | during 48 hours following surgery and after 7 days
The efficacy of pain management during 4 days past surgery | during 4 days past surgery
  Pain sensation will be assessed using the VAS scale

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek Medical Center, Afula, Israel

REFERENCES:
- [Derived] Yefet E, Nassar S, Carmeli J, Massalha M, Hasanein J, Zafran N, Rudin M, Nachum Z. Oral analgesia in fixed-time interval administration versus spinal morphine for post-Cesarean pain: a randomised controlled trial. Arch Gynecol Obstet. 2022 Apr;305(4):893-901. doi: 10.1007/s00404-021-06196-3. Epub 2021 Aug 31. PMID 34463805